CLINICAL TRIAL: NCT06276075
Title: The Influence of Therapy Enriched With the Erigo®Pro Table and Motor Imagery on the Body Balance of Patients After Stroke - a Randomized Observational Study.
Brief Title: The Impact of Erigo®Pro Therapy and Motor Imagery on the Balance of Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anna Olczak (Other)
Responsible Party: Sponsor-Investigator, Anna Olczak, PhD; Senior Specjalist of the Rehabilitation Clinic, Military Institute od Medicine National Research Institute
Organization: Military Institute od Medicine National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10/KRN/2020
Record Dates: First submitted 2024-02-18; First posted 2024-02-23 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: stroke,; motor imaging,; Erigo®Pro tilt table,; balance,; physiotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional rehabilitation (Experimental): patients performed daily physiotherapy, which included intensive preparatory training for standing and sitting positions, strengthening exercises, weight-bearing exercises, and balance and coordination exercises (from 40 to 60 minutes of therapy).
  Interventions: Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery
- Erigo®Pro (Experimental): effective therapy included 1 session on a tilting table at an angle of 42° for 20 minutes, 5 times a week (Monday to Friday) at a speed of 32 steps per minute, followed by a physiotherapy session for two weeks.
  Interventions: Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery
- motor imagery (MI) (Experimental): in addition to conventional physiotherapy, activity imagery during passive walking on the Erigo®Pro table was introduced. During the exercises on the table, the patients wore headphones that blocked out any external sounds, closed their eyes and their task was to imagine the sensation of their body moving (first-person imagination), differentiating the idea of walking in various real environments (park, forest, beach, snow, streets). in the city, walking at different speeds, going up and down stairs, running, etc.)
  Interventions: Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery

INTERVENTIONS:
Procedure: Conventional rehabilitation, the Erigo®Pro table, motor imagery — 66 stroke patients were randomly assigned to three groups (22 people each) with different therapy (conventional, with the addition of Erigo®Pro and enriched with motor imagery). The therapy duration was two weeks. Patients underwent assessment before and after completion of therapy. The study used the Trunk Stability Test, Berg Balance Scale to assess balance, as well as the Riablo device to measure static balance. Additionally, an evaluation of the superficial tension of the transverse abdominis and multifidus muscles was conducted.

SUMMARY:
The aim of the study is to examine the impact of motor imagery, Erigo®Pro tilt table intervention, and classic rehabilitation on the balance of people after a stroke.

DETAILED DESCRIPTION:
DESIGN: randomized observational study. SETTING: A hospital Rehabilitation Department. POPULATION: Sixty-six post-stroke patients mean, 64.85 ± 18.62 years. METHODS: 66 stroke patients were randomly assigned to three groups (22 people each) with different therapies (conventional, with the addition of Erigo®Pro and enriched with motor imagery). The therapy duration was two weeks. Patients underwent assessment before and after completion of therapy. The study used the Trunk Stability Test, Berg Balance Scale to assess balance, as well as the Riablo device to measure static balance. Additionally, an evaluation of the superficial tension of the transverse abdominis and multifidus muscles was conducted.

ELIGIBILITY:
Inclusion Criteria:

1) patients 6-8 weeks post-stroke, 2) aged 38-85 years, mean, 3) males and females, 4) walking with or without assistance (modified Rankin scale = 3), 5) with slight neurological deficits (NIHSS ≤7).

Exclusion Criteria:

1) stroke up to six weeks after the episode, 2) epilepsy, 3) no possibility to sit and stand, 4) persistent deficit of speech and cognitive functions, lack of attention, 5) visual disturbances, 6) depression, 7) high or very low blood pressure, dizziness, malaise.

Ages: 38 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Trunk Control Test | two weeks
  Assessment of trunk stability before and after therapy
Berg Balance Scale | two weeks
  Assessment of body balance before and after therapy
RiabloTM device | two weeks
  Assessment of static balance in the frontal plane before and after therapy
RiabloTM device | two weeks
  Assessment of static balance in the sagittal plane before and after therapy
Luna EMG | two weeks
  Assessment of the surface tension of the transverse abdominis muscle
Luna EMG | two weeks
  Assessment of the surface tension of the multifidus muscle

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Olczak, PhD, Principal Investigator — Military Institute of Medicine, Rehabilitation Clinic
Locations (1):
- Military Institute of Medicine, Warsaw, Masovian District, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olczak A, Carvalho R, Stepien A, Mroz J. The Influence of Therapy Enriched with the Erigo(R)Pro Table and Motor Imagery on the Body Balance of Patients After Stroke-A Randomized Observational Study. Brain Sci. 2025 Mar 5;15(3):275. doi: 10.3390/brainsci15030275. PMID 40149796